CLINICAL TRIAL: NCT02483806
Title: Effects of Positive End-Expiratory Pressure on Biventricular Function During One-Lung Ventilation: a Randomized Crossover Study
Brief Title: Effects of Positive End-Expiratory Pressure on Biventricular Function During One-Lung Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 4-2015-0325
Record Dates: First submitted 2015-06-19; First posted 2015-06-29 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- PEEP 0 cmH2O (Experimental): PEEP 0 cmH2O (zero end expiratory pressure, ZEEP)
  Interventions: Procedure: PEEP
- PEEP 5 cmH2O (Experimental)
  Interventions: Procedure: PEEP
- EEP 10 cmH2O (Experimental)
  Interventions: Procedure: PEEP

INTERVENTIONS:
Procedure: PEEP — After induction of anesthesia, including insertion of TEE probe, change position from supine to lateral position. Measure ABGA and cardiac indices for the baseline value. Apply each PEEP (0, 5, 10 cmH2O) serially at the random order. 6 sequences (0->5->10, 0->10->5, 5->10->0, 5->0->10, 10->5->0, 10->0->5) are equally applied to 6 patients (total 6x6=36 patients) who agreed to this study. Measure ABGA and cardiac indices after 20 min at each step of peep apply(3 times).
  Other Names: Positive EndExpiratory Pressure breathing(PEEP)

SUMMARY:
One lung ventilation (OLV) is essential during thoracic surgery. During OLV, intrapulmonary shunt can be increased resulting hypoxemia. Wang et al measured intrapulmonary shunt by transesophageal echocardiography. Although OLV technique had been advanced so far, hypoxemia during OLV reaches about 10% in spite of inspired oxygen fraction 100%. Applying PEEP(Positive End-expiratory Pressure) at dependent lung and CPAP at non-dependent lung can mitigate the hypoxemia. Above all, PEEP can be easily applicable. However, there are controversial studies whether it is supportive or not. In this prospective, cross-over study, the investigators are planning to investigate the effects of PEEP on intrapulmonary shunt, oxygenation and cardiac function as well.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for VATS lobectomy
* 40 ≤ age ≤ 80
* American Society of Anaesthesiologists(ASA) physical status classification I~III

Exclusion Criteria:

* American Society of Anaesthesiologists(ASA) physical status classification IV
* NYHA class III~IV
* Severe obstructive lung disease and/or restrictive lung disease patients
* those with end-organ diseases (i.e. heart failure, respiratory failure, hepatic failure, renal failure)
* arrhythmia
* esophageal varix
* pregnant women

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2016-05-25 (Actual); Study Completion 2016-05-25 (Actual)

PRIMARY OUTCOMES:
the effect of differential PEEP (0, 5, 10 cmH2O) by PaO2(P/F ratio) | 20 minutes after each PEEP apply
Cardiac function | 20 minutes after each PEEP apply
  cardiac function : Tei index

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Pain Medicine, Anaesthesia and Pain Research Institute, Yonsei University College of Medicine, Seoul, South Korea